CLINICAL TRIAL: NCT02303613
Title: A Validation of Current Hospital Triage Performance System Versus RETTS and Identify Trauma Patient Outcome at Moi Teaching and Referral Hospital, Kenya.
Brief Title: A Validation of Current Hospital Triage Performance System Versus RETTS
Acronym: HTPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Maria Lampi, RN, MSc DM, PhD-candidate, University Hospital, Linkoeping
Other Study IDs: KMC-001
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Wound and Injuries; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Mapping — Mapping of current triage situation regarding 30 days mortality

SUMMARY:
Background: Triage in the emergency department (ED) together with initial assessment is used to identify patient's level of urgency and treatment based on their triage level. Triage in the ED is a complex decision-making process, and several triage scales have been designed as decision support systems to guide the triage nurse to a correct decision. Worldwide there are four well known five-level triage systems in use. In 2010, 97% of all EDs in Sweden introduced a process-oriented triage scale with physiological parameters called Rapid Emergency Traige and Treatment System (RETTS). RETTS has two main assessment variables: vital signs and chief complaints, which describe the incident or symptoms that caused the patient to seek care. These two variables are evaluated and results in a color coded 5-level scale. Each level of priority has a defined time limit within which evaluation by a doctor should begin. Although, all international triage system guidelines seem to function well in western countries, they are difficult to implement and have a high failure rate in developing low-income countries. One of the reasons may be the lack of extensive training. Teaching and assessing abilities in performing mass casualty triage in inherently challenging due to the inability to accurately replicate a given disaster environment in a comprehensive way. Disaster drills and simulation exercises are ways of training triage performance and there are different tools available. One tool that can contribute to this kind of training may be the Emergo Train System® (ETS). ETS or similar interactive educational simulation systems could be used to test and evaluate incident and command systems, surge capacity, hospital preparedness and triage.

Study objective study III: The aim of the study is to validate the currently practiced system for triage in the ED in Moi Teaching and Referral Hospital in Eldoret, Kenya with RETTS. Furthermore map the current patient outcome of trauma patients.

DETAILED DESCRIPTION:
A tool has been developed by the research group. It has been developed in which on identification of trauma patient record, details will be entered and later transferred to an Excel format for ease of analysis.

Trauma patient card record for collecting data including respiratory rate, pulse, blood pressure, GCS, SaO2, body temperature, type of injury and mechanism of injury is developed will be used. Time of accident and arrival to ED, sex, age and intervention at ED will also be registered. Time at ED, number of days and where the patient has been treated during the hospital visit are also going to be registered. According to the protocol there is also a discharge evaluation where The International Classification of Disease (ICD) and Injury Severity Score (ISS) will be registered.

ELIGIBILITY:
Inclusion Criteria:

Close to 600 trauma patients of ages 14 and above seen at the ED will be captured. All patients presenting through the ED will be identified and those who meet the inclusion criteria will be recruited into the study on a daily basis until close to the 600 patient records is achieved. Patients will be followed through the ED to the receiving facilities (wards, ICU, HDU, theatre etc) -

Exclusion Criteria:

Those brought in dead, those below 14 years, revisits, or referred patients will be excluded The patient records will be traced for the entire period the patient is in the hospital or until key decisions are made on triage category by the ED or receiving units.

There may be need to follow up patients for longer but since the study has a limited period, records will have to be made up to 30 days admission for those admitted during the last month.

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Close to 600 trauma patients of ages 14 and above seen at the ED will be captured. All patients presenting through the ED will be identified and those who meet the inclusion criteria will be recruited into the study on a daily basis until close to the 600 patient records is achieved. Patients will be followed through the ED to the receiving facilities (wards, ICU, HDU, theatre etc)
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Identify and mapping of the current 30 days mortality and morbidity. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lampi, PhD-cand, Principal Investigator — Linkoeping University
Locations (1):
- Moi Teaching and Referral Hospital, Kenya., Eldoret, Kenya

REFERENCES:
- [Derived] Lampi M, Junker JPE, Tabu JS, Berggren P, Jonson CO, Wladis A. Potential benefits of triage for the trauma patient in a Kenyan emergency department. BMC Emerg Med. 2018 Nov 29;18(1):49. doi: 10.1186/s12873-018-0200-7. PMID 30497397